CLINICAL TRIAL: NCT04628130
Title: Efficacy of Yoga Based Self-Management Program for Chronic Pain: Community Based Clinical Efficacy Study
Brief Title: Efficacy of Yoga Based Self-Management Program for Chronic Pain
Status: Completed | Type: Observational
Sponsor: Aarogyam UK (Other)
Collaborators: Patanjali Yog Peeth (UK) Trust (Unknown)
Responsible Party: Sponsor
Other Study IDs: AU0211
Record Dates: First submitted 2020-11-09; First posted 2020-11-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Yoga

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Yoga Therapy — Yoga based self managed practices personalised to chronic pain patients

SUMMARY:
Chronic pain is a major health issue with substantial economic burden.To support chronic pain patients during the COVID-19 pandemic, yoga based self-managed intervention was delivered through tele-health platform. Project was designed as community-based program, creating new social networks for patients, health care providers and academics. Platform to deliver intervention and data collection was AiM COVID mobile app.

Our objective was to determine the efficacy of Yoga based self-management intervention for people living with chronic pain pain intensity, disability and health related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Chronic pain for at least 3 months
* Having access to internet and video calls

Exclusion Criteria:

* Pregnant or breast-feeding women,
* Patients not willing to give written consent
* Patients with severe psychiatric or personality disorder
* Malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community based project in partnership with community organisation, health care providers and academic included chronic pain patients for yoga self management therapy.
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2020-09-17 (Actual); Primary Completion 2020-11-05 (Actual); Study Completion 2020-11-09 (Actual)

PRIMARY OUTCOMES:
Pain intensity and disability | From baseline to 6 week post intervention
  Pain intensity and related disability was measured through Brief Pain Inventory
Health Related Quality of Life | From baseline to 6 week post intervention
  Quality of life was measured through 36-Item Short-Form Survey
Self-efficacy of pain | From baseline to 6 week post intervention
  Self efficacy was measure through Pain Self-Efficacy Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Neha Sharma, Principal Investigator — Aarogyam UK; Deepa Modi, Study Chair — East Park Medical Centre, NHS trust, Leicester; Vishwesh Kulkarni, Study Director — University of Warwick; Sunita Poddar, Principal Investigator — Patanjali Yog Peeth (UK) Trust
Locations (2):
- United Kingdom (2):
  - Aarogyam UK, Leicester, Leicestershire
  - Patanjali Yog Peeth (UK) Trust, Glasgow, Scotland

IPD SHARING:
Plan to Share IPD: Undecided